CLINICAL TRIAL: NCT04723719
Title: SIESTA Sleep IntervEntion as Symptom Treatment for ADHD - Blended CBT Sleep Intervention to Improve Sleep, ADHD Symptoms and Related Problems in Adolescents With ADHD
Brief Title: Sleep IntervEntion as Symptom Treatment for ADHD
Acronym: SIESTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Research Foundation Flanders (Other); KU Leuven (Other)
Responsible Party: Principal Investigator, Saskia Van der Oord, Prof. Dr., KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UZ Leuven
Record Dates: First submitted 2021-01-12; First posted 2021-01-26 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: ADHD; Sleep; Adolescents; CBT
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial with training group and control group.
Who Masked: Investigator
Masking Description: Stratified permuted block randomization, controlling for ADHD medication use (yes/no), is done by a masked/independent researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIESTA training + treatment as usual for ADHD (Experimental): We developed a cognitive behavioral therapy for sleep problems in adolescents with ADHD. This includes seven individual sessions with the adolescent and two individual sessions with the parent(s)/guardian(s). Participants receive this CBT training called SIESTA next to their treatment as usual for ADHD symptomatology (mostly ADHD-medication).
  Interventions: Behavioral: SIESTA; Other: Treatment as usual for ADHD
- Treatment as usual for ADHD only (Active Comparator): Participants continue their treatment as usual for ADHD (mostly ADHD-medication).
  Interventions: Other: Treatment as usual for ADHD

INTERVENTIONS:
Behavioral: SIESTA — SIESTA is a CBT sleep training for adolescents with ADHD with a focus on sleep hygiene, motivational interviewing and planning and organization.
  Other Names: Sleep IntervEntion as Symptom Treatment for ADHD
  Arms: SIESTA training + treatment as usual for ADHD
Other: Treatment as usual for ADHD — Participants continue their treatment as usual for ADHD.
  Other Names: TAU

SUMMARY:
Up to 72% of adolescents with ADHD portray sleep problems. The most common sleep difficulties in adolescents with ADHD are initial insomnia, nocturnal awakenings, non-restorative or restless sleep. These difficulties seem to be causally related to increased ADHD symptom impairment, oppositional and depressive symptomatology, and functional impairments in daily life, resulting in a vicious circle of sleep problems and impairment. Thus, reducing sleep problems is an important intervention target. However, to date there is no evidence-based cognitive behavioral sleep treatment available. Sleep-focused treatments need adaptation towards this developmental phase/disorder for effectiveness, as ADHD and sleep problems are bi-directional. Therefore, a blended treatment targeting the core deficits integrating motivational interviewing, planning skills and sleep interventions is needed. Thus, the aim of this project is testing the short and 3 months follow-up effectiveness of the blended CBT sleep intervention in adolescents with ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Attending secondary education and between 13-17 years old
2. prior diagnosis of ADHD (any presentation) and confirmation of DSM-5 criteria of ADHD in current study
3. Displaying sleep problems for at least 3 nights per week for at least 3 months

   1. sleep onset latency of at least 20-30 minutes
   2. and/or wake after sleep onset greater than 30 min
   3. and/or an average sleep time of less than 7 hours
   4. and at least one poor sleep hygiene practice
   5. and experienced distress as indicated by parent/guardian and/or adolescent.
4. estimated IQ≥80
5. stable ADHD medication use at least 4 weeks before start of treatment and no dose or medication type changes planned during active treatment

Exclusion Criteria:

1. the following comorbidities: sleep-breathing disorder, restless leg syndrome, narcolepsy, conduct disorder, depressive disorder with suicide risk or active suicidality, autism spectrum disorder, or substance use disorder, with an exception for nicotine
2. acute crisis situation at home
3. physical problems that interfere with sleep (e.g. pain) or medical disorders and related medication that could affect sleep
4. participation in a behaviorally based sleep intervention in the 6 months prior to our study
5. currently taking pharmacological medication for sleep (including melatonin), anxiety or depression. Participation will be allowed after a two-week wash-out period of the medication

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Sleep architecture objective TST pre-test to post-test | From pre-test to post-test (+- 8 weeks)
  objective (actigraphy) sleep architecture (specified as TST in hours and minutes)
Sleep architecture objective SOL pre-test to post-test | From pre-test to post-test (+- 8 weeks)
  objective (actigraphy) sleep architecture (specified as SOL in hours and minutes)
Sleep architecture objective SE pre-test to post-test | From pre-test to post-test (+- 8 weeks)
  objective (actigraphy) sleep architecture (specified as SE = TST/time in bed in percentage)
Sleep architecture objective NoA pre-test to post-test | From pre-test to post-test (+- 8 weeks)
  objective (actigraphy) sleep architecture (specified as NoA)
Sleep architecture subjective TST pre-test to post-test | From pre-test to post-test (+- 8 weeks)
  subjective (sleep logs) sleep architecture (specified as TST in hours and minutes)
Sleep architecture subjective SOL pre-test to post-test | From pre-test to post-test (+- 8 weeks)
  subjective (sleep logs) sleep architecture (specified as SOL in hours and minutes)
Sleep architecture subjective SE pre-test to post-test | From pre-test to post-test (+- 8 weeks)
  subjective (sleep logs) sleep architecture (specified as SE = TST/time in bed in percentage)
Sleep architecture subjective NoA pre-test to post-test | From pre-test to post-test (+- 8 weeks)
  subjective (sleep logs) sleep architecture (specified as NoA)
Sleep architecture objective TST pre-test to follow-up | From pre-test to follow-up (+-3 months after posttest)
  objective (actigraphy) sleep architecture (specified as TST in hours and minutes)
Sleep architecture objective SOL pre-test to follow-up | From pre-test to follow-up (+-3 months after posttest)
  objective (actigraphy) sleep architecture (specified as SOL in hours and minutes)
Sleep architecture objective SE pre-test to follow-up | From pre-test to follow-up (+-3 months after posttest)
  objective (actigraphy) sleep architecture (specified as SE = TST/time in bed in percentage)
Sleep architecture objective NoA pre-test to follow-up | From pre-test to follow-up (+-3 months after posttest)
  objective (actigraphy) sleep architecture (specified as NoA)
Sleep architecture subjective TST pre-test to follow-up | From pre-test to follow-up (+-3 months after posttest)
  subjective (sleep logs) sleep architecture (specified as TST in hours and minutes)
Sleep architecture subjective SOL pre-test to follow-up | From pre-test to follow-up (+-3 months after posttest)
  subjective (sleep logs) sleep architecture (specified as SOL in hours and minutes)
Sleep architecture subjective SE pre-test to follow-up | From pre-test to follow-up (+-3 months after posttest)
  subjective (sleep logs) sleep architecture (specified as SE = TST/time in bed in percentage)
Sleep architecture subjective NoA pre-test to follow-up | From pre-test to follow-up (+-3 months after posttest)
  subjective (sleep logs) sleep architecture (specified as NoA)
Sleep problems SSHS pre-test to post-test | From pre-test to post-test (+- 8 weeks)
  subjective sleep problems assessed by questionnaires (SSHS)
Sleep problems CSRQ pre-test to post-test | From pre-test to post-test (+- 8 weeks)
  subjective sleep problems assessed by questionnaires (CSRQ)
Sleep problems CSHQ pre-test to post-test | From pre-test to post-test (+- 8 weeks)
  subjective sleep problems assessed by questionnaires (CSHQ)
Sleep problems SSHS pre-test to follow-up | From pre-test to follow-up (+-3 months after posttest)
  subjective sleep problems assessed by questionnaires (SSHS)
Sleep problems CSRQ pre-test to follow-up | From pre-test to follow-up (+-3 months after posttest)
  subjective sleep problems assessed by questionnaires (CSRQ)
Sleep problems CSHQ pre-test to follow-up | From pre-test to follow-up (+-3 months after posttest)
  subjective sleep problems assessed by questionnaires (CSHQ)
Sleep hygiene pre-test to post-test | From pre-test to post-test (+- 8 weeks)
  subjective sleep hygiene assessed by questionnaires (ASHSr)
Sleep hygiene pre-test to follow-up | From pre-test to follow-up (+-3 months after posttest)
  subjective sleep hygiene assessed by questionnaires (ASHSr)

SECONDARY OUTCOMES:
ADHD symptoms pre-test to post-test | From pre-test to post-test (+- 8 weeks)
  Assessed by parents (DBDRS)
ADHD symptoms pre-test to follow-up | From pre-test to follow-up (+-3 months after posttest)
  Assessed by parents (DBDRS)
Parent-adolescent conflict pre-test to post-test | From pre-test to post-test (+- 8 weeks)
  Assessed by parents (CBQ)
Parent-adolescent conflict pre-test to follow-up | From pre-test to follow-up (+-3 months after posttest)
  Assessed by parents (CBQ)
Homework problems pre-test to post-test | From pre-test to post-test (+- 8 weeks)
  Assessed by parents (HPC)
Academic competence pre-test to post-test | From pre-test to post-test (+- 8 weeks)
  Assessed by teacher (CPS)
Homework problems pre-test to follow-up | From pre-test to follow-up (+-3 months after posttest)
  Assessed by parents (HPC)
Academic competence pre-test to follow-up | From pre-test to follow-up (+-3 months after posttest)
  Assessed by teacher (CPS)
Comorbidities: oppositional-defiant disorder pre-test to post-test | From pre-test to post-test (+- 8 weeks)
  Assessed by parents (DBDRS)
Comorbidities: anxiety pre-test to post-test | From pre-test to post-test (+- 8 weeks)
  Assessed by adolescent (SCARED-R)
Comorbidities: depression pre-test to post-test | From pre-test to post-test (+- 8 weeks)
  Assessed by adolescent (CDI-2)
Comorbidities: oppositional-defiant disorder pre-test to follow-up | From pre-test to follow-up (+-3 months after posttest)
  Assessed by parents (DBDRS)
Comorbidities: anxiety pre-test to follow-up | From pre-test to follow-up (+-3 months after posttest)
  Assessed by adolescent (SCARED-R)
Comorbidities: depression pre-test to follow-up | From pre-test to follow-up (+-3 months after posttest)
  Assessed by adolescent (CDI-2)

CONTACTS AND LOCATIONS:
Overall Officials: Saskia Van der Oord, PhD, Principal Investigator — KU Leuven
Locations (1):
- UPC Leuven, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After all waves of the study are finished and data analyzed. This is expected to happen in 2024. Data will be available 25 years after the study.

REFERENCES:
- [Derived] Keuppens L, Marten F, Baeyens D, Boyer B, Danckaerts M, van der Oord S. Sleep IntervEntion as Symptom Treatment for ADHD (SIESTA)-Blended CBT sleep intervention to improve sleep, ADHD symptoms and related problems in adolescents with ADHD: Protocol for a randomised controlled trial. BMJ Open. 2023 Apr 13;13(4):e065355. doi: 10.1136/bmjopen-2022-065355. PMID 37055205